CLINICAL TRIAL: NCT00551668
Title: A Prospective, Randomized Study of Operative and Nonoperative Treatment for Primary Traumatic Patellar Dislocation in Young Adults With a Median 7-Year Follow-Up
Brief Title: A Prospective, Randomized Study of Operative and Nonoperative Treatment for Primary Traumatic Patellar Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Defense Forces (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R1199/8.1/D/II
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Patellar Dislocation
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Operative
  Interventions: Procedure: proximal patellar surgery
- 2 (Experimental): Nonoperative
  Interventions: Procedure: Nonoperative

INTERVENTIONS:
Procedure: proximal patellar surgery — Initial proximal patellar surgery
  Arms: 1
Procedure: Nonoperative — Nonoperative without surgery
  Arms: 2

SUMMARY:
The objective of this prospective, randomized cohort study was to evaluate the clinical results between operative and nonoperative treatment of primary patellar dislocation.

DETAILED DESCRIPTION:
There is no consensus about management of acute traumatic primary patellar dislocations in young physically active adults. Acute lateral patellar dislocation is a relatively common injury among young adults. Proper treatment for this condition has been researched for decades. However, there is a lack of prospective randomized studies to evaluate the different treatment options for traumatic primary patellar dislocations. Therefore a prospective, randomized study was designed with the aim to compare the outcome of operative versus nonoperative treatment of primary traumatic patellar dislocations in young adults.

ELIGIBILITY:
Inclusion Criteria:

* An acute primary traumatic patellar dislocation

Exclusion Criteria:

* Previous dislocation or subluxation of the patella
* Pre-existing ipsilateral or contralateral knee pathology
* Previous knee trauma or patellar fracture.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-01; Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Number of redislocations | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Harri Pihlajamäki, M.D., Ph.D., Study Director — Centre for Military Medicine, Lahti, Finland